CLINICAL TRIAL: NCT02010359
Title: Omega-3 PUFA Suppress Adipochemokines
Brief Title: Fish Oils and Adipose Inflammation Reduction
Acronym: FAIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1K23DK095913-01A1 (NIH); 1K23DK095913-01A1 (NIH)
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lovaza (Experimental): Lovaza 4 grams daily (2 1-gram capsules twice daily) will be given for 8 weeks
  Interventions: Drug: Lovaza
- Placebo (Placebo Comparator): An inactive Placebo (2 pills twice daily) will be given for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lovaza — Lovaza 4 grams per day
  Arms: Lovaza
Drug: Placebo — Placebo pill
  Arms: Placebo

SUMMARY:
This study is a clinical trial designed to assess whether fish oil treatments are effective in the prevention of obesity-related fat tissue (adipose) inflammation. Specifically it addresses the hypothesis that fish oils treatments will reduce signaling by chemokine pathways (fractalkine and MCP-1) important in adipose tissue for the recruitment and activation of certain white blood cells (macrophages). The study is a double-blind placebo-controlled trial of the fish oil Lovaza from GlaxoSmithKline (omega-3-acid ethyl esters; a combination of ethyl esters of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA)) in obese non-diabetic adults, to determine if Lovaza decreases markers of inflammation and macrophage activation in adipose and blood and understand the mechanism by which fish oils affect inflammation.

DETAILED DESCRIPTION:
We propose to conduct a parallel arm, double blind, placebo-controlled trial to understand the anti-inflammatory and metabolic effects of marine derived omega-3 fatty acids (EPA + DHA) on obesity-related inflammation and chemokine signaling in humans. Obese (BMI>30 kg/m2) but non-diabetic young males and females (n~44; 25 to 50 years of age) taking no omega-3 fatty acid (EPA + DHA) supplements and consuming a low fish diet (defined as usual intake of high omega-3 fish (tuna and other non-fried fish) < 3 to 4 servings per month) will be included. A low habitual fish intake is important to control EPA + DHA intake during the supplement period (see exclusion criteria below). Subjects also will be required to maintain their current fish intake throughout the treatment period.

There will be two treatment groups; (1) placebo and (2) omega-3 fatty acids 4 grams/day. The trial will be randomized, double blind, placebo-controlled, with parallel treatment groups; treatment with omega-3 fatty acids 8 weeks. We will enroll participants until at least 22 subjects per study-arm complete all study visits (i.e., at least 44 participants).

Prescription Lovaza (omega-3-acid ethyl esters) from GlaxoSmithKline at 4 grams day (2 1-gram capsules twice daily, with food) will be used. We expect this dose to be safe because it is a dose that is recommended, and routinely used, for management of moderate or worse hypertriglyceridemia (levels > 400 mg/dL). We will use matching placebo capsules so that all participants are taking 2 capsules twice daily - with food as recommended in clinical practice.

The study duration was chosen in order to provide adequate time for potential anti-inflammatory effects of treatments without requiring maximum lipid modifying effects while also reducing the potential for drop-out and loss to follow up that is associated with longer study durations.

Participants will be recruited from the Preventive Cardiology Research databases, comprised of healthy subjects who have participated in previous research studies and who have asked to be contacted for future studies. Potential participants will also be recruited via local IRB-approved flyers, internet, and newspaper advertisements (see flyer and advertisement attached) targeting the Delaware Valley region.

STUDY PROCEDURES

Informed Consent Before study initiation, the clinical protocol, the Informed Consent Form (ICF), and any advertisements for subject recruitment will be submitted for review and approval to the Institutional Review Board (IRB). The investigator, or his designated research staff, will obtain written informed consent from each subject enrolled in the study, in accordance with the U.S. Food and Drug Administration (FDA) regulations 21 CFR parts 50.20-50.27. It is the responsibility of the investigator to ensure that informed consent is obtained from the subject or his/her guardian or legal representative before any activity or treatment is undertaken which is not part of routine care.

Safety Assessments Safety will be evaluated by the incidence, severity, and relationship to treatment agent of adverse events.

Monitoring for Adverse Events: Details of all AEs that occur after the first dose of study drug will be collected as indicated in Section 12. Any illness or injury that occurs before the first dose of a study drug will be recorded under Medical History and evaluated to determine if the occurrence affects the patient's eligibility to participate in the study. Subjects will be asked the following standard questions by the designated clinical evaluator: At clinic check-ins:

1. "Have you had any medical problems since your last visit?"
2. "Have any medical problems present at your last visit changed, i.e., stopped, worsened, or improved?"
3. "Have you taken any medicines, other than study drug, since your last visit?" Any spontaneous AE information provided by the patient will be recorded. NOTE: An AE may be a new disease(s), any untoward event(s), or an exacerbation of a pre existing condition. See Section 12.0 for complete details.

Adipose biopsy: Approximately 500-1000 mg of subcutaneous adipose tissue will be biopsied from the gluteal region, processed, weighed and frozen until analyzed. Adipose tissue will be obtained through a small (~5mm) incision under local anesthesia (2% Lidocaine without epinephrine), as has been previously described13-15. A portion (200 mg) of the samples will be flash frozen and analyzed for gene expression and protein assays. Another portion (500-800 mg) will be placed in sterile media and undergo digestion with collagenase, filtration, and centrifugation for separation of the stromal vascular fraction (SVF). SVF cells will be stained with antibodies for flow cytometer analysis. Finally, remaining tissue will be fixed in paraffin for immunohistochemistry.

6.5 Subgingival analysis

Saliva samples will be collected using the OMNIgene DISCOVER (OM-505) kit (DNA Genotek), an all-in-one kit which collects and stabilizes both microbial DNA and RNA in saliva. Samples will be stored at -80C prior to extraction. Nucleic acids will be extracted using the QIAGEN QIAamp MinElute Virus Spin Kit (Qiagen). Subgingival plaque samples will be obtained from 3 oral cavity regions in each subject (2 samples per region) using a soft-bristled microbrush (DenTek). Specimens will be collected from the same anatomical location in all subjects. DNA will be isolated using the PSP Spin Stool DNA kit (Invitec). DNA samples will be amplified using V1-V2 region primers targeting bacterial 16S genes and sequenced using IlluminaHiSeq or 454 Pyrosequencing technology.

Specific Study Procedures (by visit)

Screening (Visit 1) Potential participants will be screened first by a telephone or e-mail interview with the research coordinator (see Appendix B for email interview form; for telephone interviews this information will be verbally exchanged). Participants who meet initial study requirements will be invited for a screening visit (visit 1) at the CTRC. Prior to this visit, participants will receive a detailed health questionnaire (see Appendix C) that has been used in numerous previous studies that addresses questions regarding past medical history, current use of medications and dietary supplements, exercise and social habits. In addition, participants will be asked about fish consumption in order to ensure recruitment of subjects with lower EPA + DHA intake during the study period. Participants will be asked to complete these questionnaires at home and bring the completed forms with them to their screening visit. During the screening visit, they will meet with research staff to review and sign an IRB-approved consent form. Research staff will review the health questionnaire with the participant as well as measure weight, height, waist and hip circumference, sitting blood pressure and heart rate. A brief physical exam will be performed as well as an electrocardiogram (ECG). In addition, participants will have blood drawn (after a 12 hour fast) for evaluating fasting lipids, glucose, serum chemistries and liver function and a complete blood count. Female participants will also be asked to provide a urine sample for a pregnancy test. These laboratory parameters are included to assure the participant meets eligibility criteria and that he/she is generally in good health. Once all clinical data has been reviewed, study personnel will contact each study volunteer to let them know if they are eligible.

Randomization visit (Visit 2) One to four weeks after the screening Visit 1, eligible participants will return to the CTRC after a 12 hour fast for a 2 hour visit. Participants will be asked to brush their teeth after their last meal the day before the visit, or at the start of the 12-hour fasting period, and to refrain from additional brushing or use of mouthwash until after the study visit. Participants will meet with a research nurse / coordinator who will assess any change in medical history and medication use, as well as review any adverse events. Blood pressure, heart rate, height and weight will be measured, blood and urine will be collected for pre-randomization baseline efficacy measures and a urine pregnancy test performed for all females. The simple fish consumption questionnaire will be administered to assess any changes to the level of omega-3 intake in the diet.

They will also be asked to record all food and beverages consumed on dietary records on 3 days prior to the visit, as well as completing a digestive health questionnaire and diet history questionnaire. All nutrient data collected from 3-day dietary records will be analyzed by Food Processor 8.1 (06/03, Escha). Participants will be asked to complete these questionnaires at home and bring the completed forms with them to their study visit. If a subject is unable to print out or complete the forms at home, they will be completed at the visit.

Saliva and subgingival plaque samples will be taken for assessment of oral microbiome. Saliva samples will be collected using a standardized kit. Under the supervision of study personnel, subjects will be given the kit, which consists of a funnel attached to a tube, and instructed to spit into the funnel until the amount of liquid reaches a fill line located on the outside of the attached tube. Once the proper amount has been collected, the lid of the funnel will be closed and the funnel removed from the tube. The tube is then capped and shaken for about 10 seconds. Subgingival plaque samples will be collected by swabbing several regions of the buccal mucosa using microbrushes. A separate brush will be used for each swab and two samples will be collected from each region.

In order to establish effects of treatments on adipose inflammatory parameters, we will obtain gluteal region subcutaneous adipose tissue biopsies under local anesthesia (2% Lidocaine). A detailed description of the adipose collection procedures is given in Section 6.4. Participants will then be randomized to drug or placebo group. Supplies of study drug will be provided to last 8 weeks (4 pills/day of either Lovaza or placebo).

Participants will be provided verbal and written instruction to take the study drugs as follows; 2 fish oil/placebo with food in the morning, 2 fish oil/placebo with food in the evening. A pill diary will be given to all subjects.

Telephone / E-mail Follow up (Visit 3) Participants will be contacted by telephone or e-mail approximately four weeks (visit 3) post-randomization to review medication compliance and pill diary, adverse events and any changes in fish consumption. Participants with <80% apparent adherence to study medication will be counseled to increase compliance so that their adherence at 8 weeks will be ≥80%.

Completion Visit (Visit 4) Participants will come to the CTRC after a 12 hour fast. Participants will meet with a study coordinator who will assess changes to the medical history and medication use. They will also be asked to record all food and beverages consumed on dietary records on 3 days prior to the visit. Any adverse events will be recorded, pill diary reviewed, and study medications will be counted (pill count) Weight and height will be recorded and BMI calculated. ECG will be performed. Blood will be drawn for post-drug screening of liver functions and chemistries as well as for all outcome-related measures (lipids, insulin/glucose, inflammatory markers). Urine for efficacy measures will also be collected. Urine pregnancy test will be performed in all females. Saliva and subgingival plaque samples will be taken to assess for any change in oral microbiome by the treatment. An adipose biopsy will be performed as above.

ELIGIBILITY:
Inclusion Criteria:

1. Men and non-pregnant/lactating women between the ages of 25 and 50.
2. Body Mass Index (BMI) ≥30 kg/m2
3. Participants who are able to give written informed consent and willing to comply with all study-related procedures.

Exclusion Criteria:

1. Diabetes Mellitus (glucose fasting >126, or random >200, Hemoglobin A1C>6.5 %, or use of any anti-diabetic agent)
2. Self-reported fish or shellfish allergy
3. Planned usage of any prescription or non-prescription medication (other than contraceptive pills or devices) during the study period.
4. Recent (within 6 months) use of fish oil supplements or self- reported dietary intake of >3 servings of fish/month
5. Blood pressure >140/90
6. Recent (within 6 months) use of statins, niacin, or fenofibrates
7. Current or planned pregnancy/lactation. Pre-menopausal women unwilling to prevent pregnancy by use of the following approved contraceptive strategies: diaphragm, cervical cap, condom with spermicide, surgical sterility, birth control pills, Depo-Provera injection, Intra-uterine device, progestin implant, or abstinence.
8. History of liver disease or abnormal liver function tests (aspartate aminotransferase, Alanine transaminase, Alkaline Phosphatase, gamma-glutamyl transpeptidase > 1.5x Upper Limit normal; bilirubin > 2x upper limit normal) at Screening Visit
9. Men who are unwilling to limit alcohol consumption to < 14 alcoholic drinks per week or < 4 alcoholic drinks per occasion while participating in the study
10. Women who are unwilling to limit alcohol consumption to < 7 alcoholic drinks per week or < 3 alcoholic drinks per occasion while participating in the study.
11. Hemoglobin less than 11.0 g/dL
12. Any reported arrhythmia, usage of anti-arrhythmic therapy, or abnormal screening electrocardiogram
13. Known bleeding disorder or coagulopathy
14. Any major active rheumatologic, pulmonary, hematologic or dermatologic disease or inflammatory condition or minor active infection
15. Self-reported history of HIV positive
16. Patients who have undergone any organ transplant
17. Individuals who currently use tobacco products or have done so in the previous 30 days
18. Treatment with aspirin, non steroidal anti-inflammatories, COX-2 inhibitors, steroids or any immunomodulatory therapy 2 weeks prior to the Screening Visit
19. Participants who are unwilling to eliminate omega-3 fatty acid (EPA + DHA) supplements and/or fortified food, or have their usual intake of high omega-3 fish (tuna and other non-fried fish) be > 3 to 4 servings per month as assessed by a simple screening questionnaire
20. Recent (within 6 months) treatment with coumarin-type anticoagulants
21. Positive urine pregnancy test result.
22. Self-reported history of injected recreational drug use.
23. Any medical condition or abnormal laboratory value that is judged clinically significant by an investigator

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2014-06; Primary Completion 2017-06 (Actual); Study Completion 2017-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachana Shah, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Shah RD, Tang ZZ, Chen G, Huang S, Ferguson JF. Soy food intake associates with changes in the metabolome and reduced blood pressure in a gut microbiota dependent manner. Nutr Metab Cardiovasc Dis. 2020 Aug 28;30(9):1500-1511. doi: 10.1016/j.numecd.2020.05.001. Epub 2020 May 18. PMID 32620337

RESULTS

PARTICIPANT FLOW:
Groups:
- Lovaza: Lovaza 4 grams daily (2 1-gram capsules twice daily) will be given for 8 weeks
  Lovaza
- Placebo: An inactive Placebo (2 pills twice daily) will be given for 8 weeks
  Placebo
Period: Overall Study
Arm/Group | Lovaza | Placebo
Started | 15 | 14
Completed | 13 | 12
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lovaza | Placebo | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (9.4) | 37.4 (8.4) | 36.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 9 | 6 | 15
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25
BMI [Mean (Standard Deviation); unit: kg/m^2] | 36.1 (5.5) | 35.9 (6.1) | 36 (5.7)
fasting glucose [Mean (Standard Deviation); unit: mg/dl] | 86.4 (11.6) | 87.8 (10.2) | 87.1 (10.4)
fasting triglyceride [Mean (Standard Deviation); unit: mg/dl] | 138.8 (107.6) | 92.9 (35.1) | 116.8 (83.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Fractalkine Levels
Description: Quantification of fractalkine levels in plasma at baseline and after 8 weeks of Lovaza or placebo will be compared.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Lovaza | Placebo
Number analyzed (Participants) | 13 | 12
ng/ml
  baseline | 0.42 (0.1) | 0.46 (0.1)
  8 weeks | 0.48 (0.1) | 0.45 (0.1)

2. Secondary Outcome: Change in Plasma Interleukin 6 (IL-6)
Description: Quantification of plasma IL-6 at baseline and after 8 weeks of Lovaza/placebo will be compared.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Lovaza | Placebo
Number analyzed (Participants) | 13 | 12
pg/ml
  baseline | 2.1 (1.6) | 1.8 (2.0)
  8 weeks | 2.0 (1.5) | 2.0 (1.9)

3. Secondary Outcome: Change in Plasma Monocyte Chemotactic Protein-1 (MCP-1)
Description: Quantification of plasma MCP-1 at baseline and after 8 weeks of Lovaza/placebo will be compared
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Lovaza | Placebo
Number analyzed (Participants) | 13 | 12
pg/ml
  baseline | 135 (15.8) | 139 (30.8)
  8 weeks | 133 (29.1) | 123 (54.1)

4. Secondary Outcome: Change in Plasma Tumor Necrosis Factor Alpha (TNFalpha)
Description: Quantification of plasma TNFalpha at baseline and after 8 weeks of Lovaza/placebo will be compared
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Lovaza | Placebo
Number analyzed (Participants) | 13 | 12
pg/ml
  baseline | 0.72 (0.51) | 0.74 (0.23)
  8 weeks | 0.76 (0.21) | 0.74 (0.13)

5. Secondary Outcome: Change in the Ratio of Circulating Monocyte Subpopulations
Description: Ratio of inflammatory CX3CR1lowCCR2+ to less inflammatory CX3CR1hiCCR2- monocytes by flow cytometry at baseline and after 8 weeks of Lovaza/placebo will be compared
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Lovaza | Placebo
Number analyzed (Participants) | 13 | 12
ratio
  baseline | 0.31 (0.11) | 0.35 (0.15)
  8 weeks | 0.25 (0.1) | 0.31 (0.05)

6. Secondary Outcome: Change in mRNA Expression of Fractalkine in Adipose
Description: relative mRNA quantification (fold change) from baseline to 8 weeks of Lovaza/placebo will be compared in each subject
Time Frame: Baseline and 8 weeks
Population: There were 4 participants that did not have sufficient adipose tissue in the biopsy for RT-PCR
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Lovaza | Placebo
Number analyzed (Participants) | 10 | 11
fold change | 1.67 (1.1) | 1.06 (0.6)

7. Secondary Outcome: Change in mRNA Levels of MCP-1 in Adipose
Description: relative mRNA quantification (fold change) from baseline to 8 weeks of treatment in Lovaza vs. placebo groups, as measured by RT-PCR
Time Frame: Baseline and 8 weeks
Population: 4 participants did not have sufficient adipose tissue in biopsy for RT-PCR
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Lovaza | Placebo
Number analyzed (Participants) | 10 | 11
fold change | 1.2 (0.7) | 1.05 (0.6)

8. Secondary Outcome: Change in mRNA Levels of IL6 in Adipose
Description: as for outcome 7
Time Frame: Baseline and 8 weeks
Population: 4 participants did not have sufficient adipose tissue from biopsy for RT PCR
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Lovaza | Placebo
Number analyzed (Participants) | 10 | 11
fold change | 0.91 (1.1) | 1.08 (2.3)

9. Secondary Outcome: Change in mRNA Levels of TNFalpha in Adipose
Description: as for outcome 7
Time Frame: Baseline and 8 weeks
Population: 4 subjects did not have sufficient adipose tissue from biopsy for RT-PCR
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Lovaza | Placebo
Number analyzed (Participants) | 10 | 11
fold change | 1.2 (3.8) | 2.5 (5.8)

10. Secondary Outcome: Change in Ratio of Adipose Tissue Macrophage Subpopulation
Description: Ratio of M1 to M2 macrophages in adipose by flow cytometry at baseline and after 8 weeks Lovaza/placebo will be compared
Time Frame: Baseline and 8 weeks
Population: 4 participants did not sufficient adipose tissue from biopsy for flow cytometry analysis
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Lovaza | Placebo
Number analyzed (Participants) | 10 | 11
ratio
  baseline | 0.52 (0.3) | 0.64 (0.42)
  8 weeks | 0.36 (0.52) | 0.42 (0.38)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Lovaza | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 2/13 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lovaza (N=13) | Placebo (N=12)
Skiing accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Knee injury during skiing during study participation
Headache (Nervous system disorders) | 1 (2) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT02010359/Prot_SAP_000.pdf